CLINICAL TRIAL: NCT05756855
Title: Young Adults With Violent Behavior During Early Psychosis: An Open Pilot Trial
Brief Title: Young Adults With Violent Behavior During Early Psychosis (Aim 2)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Paul S. Appelbaum, Elizabeth K. Dollard Professor of Psychiatry, Medicine and Law, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAU8528; K23MH126312 (NIH); NYSPI 8451 (Other: New York State Psychiatric Institute Institutional Review Board)
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Schizophreniform Disorders; Delusional Disorder; Other Specified Schizophrenia Spectrum and Other Psychotic Disorder
Keywords: psychosis; schizophrenia; violence; aggression; intervention
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid; Aggression

STUDY DESIGN:
Intervention Model Description: open pilot clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- behavioral intervention (Experimental): This will involve conducting a 12-week open pilot trial (up to n=16 dyads of EIS clinicians-EIS participants) to test the feasibility and acceptability of the adapted Psychological Interventions for Coping with Anger and Schizophrenia: a study of outcomes (PICASSO) intervention in the OnTrackNY setting.
  Interventions: Behavioral: adapted behavioral intervention

INTERVENTIONS:
Behavioral: adapted behavioral intervention — cognitive behavioral therapy based intervention that focuses on anger, violence, and psychosis
  Other Names: PICASSO

SUMMARY:
This study aims to provide an evidence-based behavioral intervention to reduce violent behavior for individuals experiencing early psychosis.

DETAILED DESCRIPTION:
The investigators will conduct an open pilot trial of a behavioral intervention to reduce violent behavior within the OnTrackNY network. The focus of this open pilot is to explore the acceptability and feasibility of the intervention. The study will enroll early intervention service (EIS) clinician - EIS participant dyads. The planned sample size is 3-4 EIS clinicians and 10-16 EIS participants (up to n=16 dyads). This real-world open pilot will provide feedback to help tailor the intervention to the OnTrackNY setting.

ELIGIBILITY:
Inclusion Criteria for EIS participants:

* Ages 16 to 30 who have experienced nonaffective psychosis with a diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, other specified/unspecified schizophrenia spectrum and other psychotic disorders (International Classification of Disease Clinical Modification (ICD-10-CM) Diagnosis Code F20.x)
* Receive First Episode Psychosis (FEP) treatment in one of OnTrackNY clinics/sites with an eligible EIS clinicians
* Willing to participate in research interviews after each study visit during the study period

Exclusion Criteria:

* Unable to provide informed consent
* Not fluent (speaking, reading, writing) in English

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean Acceptability of Intervention Measure (AIM) | 12 weeks
  The AIM is a 4-item measure of the acceptability of the intervention, to be completed by EIS clinicians. Scores range from 1-4 with higher score indicating high acceptability.
Mean Feasibility of Intervention Measure (FIM) | 12 weeks
  The FIM is a 4-item measure of the feasibility of the intervention, to be completed by EIS clinicians. Scores range from 1-4 with higher score indicating high feasibility.
Number of EIS Participants in Attendance | 12 weeks
  The number of EIS participants that attend the cognitive behavioral therapy sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Appelbaum, MD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Findings from this study will be presented to research peers, clinicians, and the public through Presentations at Scientific Meetings, Regional Research or Educational Meetings, Newsletters and Social Media and Peer-Reviewed Publications. Those events will occur during or at the conclusion of the study.
Time Frame: Descriptive and raw data will be submitted on an annual basis. Unpublished de-identified data will be shared within one year after project completion, or when the data are published, whichever is earlier.
Access Criteria: Data and materials will be made available for research to investigators working under a Federal Wide Assurance who meet security measures and data use agreement criteria associated with public repositories, including the National Database for Clinical Trials related to Mental Illness (NDCT) and the National Institute of Mental Health (NIMH) Database of Cognitive Training and Remediation Studies (DoCTRS).